CLINICAL TRIAL: NCT03093831
Title: A Phase II Investigator Sponsored Multi-Centre Trial of the Bruton's Tyrosine Kinase (BTK) Inhibitor Ibrutinib in Patients With Relapsed or Refractory Marginal Zone Lymphoma
Brief Title: Phase II Study of Ibrutinib in Patients With Relapsed or Refractory Marginal Zone Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not meet the objectives and terminated early on 17 Jul 2020 due to poor recruitment
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore General Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54179060LYM2009
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Lymphoma, B-Cell, Marginal Zone
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib (Experimental)
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — 560mg administered orally once daily.
  Other Names: PCI-32765; Imbruvica

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Ibrutinib in predominantly Asian patients with relapsed or refractory marginal zone lymphoma.

DETAILED DESCRIPTION:
Patient sample:

Patients with histologically proven marginal zone lymphoma (splenic, nodal and extra-nodal subtypes included).

Other important requirements for recruitment into the study:

* Prior treatment with one or more lines rituximab or rituximab-based chemoimmunotherapy with failure to achieve at least a partial response (PR) or documented disease progression
* Age ≥ 21 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* At least 1 measurable disease site on computed tomography (CT) scan that is at least 1.5cm in the longest dimension.
* Patient must have an indication for treatment e.g., symptoms from disease, bulky disease (>5cm), threatened end-organ function, or cytopenias requiring transfusion or growth factor support

Dosage and Dose Regimen:

560mg of Ibrutinib is administered orally once daily. Patients with mild liver impairment (Child's-Pugh A), ibrutinib 140mg (1 x 140mg capsule) will be administered instead. The patient will continue on treatment until one of the following occurs:

* Patient has disease progression (as assessed by the investigator).
* Patient has an intercurrent illness or adverse events that prevents further ibrutinib administration.
* Patient decides to withdraw from the study.
* Investigator considers withdrawal to be in the best interest of the patient.
* Patient requires continuous therapy on a prohibited concomitant medication and no alternative medications or therapies are available as a replacement to the prohibited medication.
* Patient is lost to follow-up.
* Patient is non-compliant.
* Patient becomes pregnant.
* Study termination by the Sponsor or regulatory authority.
* Death
* Completed 3 years of ibrutinib treatment

Assessment:

CT Neck to pelvis or FDG-PET/CT skull base to mid-thigh to be performed repeated after every 12 weeks

Statistical considerations:

The primary objective of this study is to determine the efficacy of ibrutinib in Asian patients with relapsed or refractory MZL. We will consider an ORR of 50% to be desirable. Simon's 2-stage minimax design will be used to test the null hypothesis that the overall response rate will be less than or equal to 20% (response rate that is considered not clinically compelling). Twelve subjects will be included in the first stage, and if there are at least 3 responders, a total of 21 subjects will be enrolled. The treatment will be declared ineffective if there are less than 8 responders in total. This design has 90% power to detect an overall response rate of 50% at a 5% significance level.

Study Endpoints:

Primary:

1. Overall response rates (complete remission [CR] + partial remission [PR])

Secondary:

1. Survival parameters

   * Progression-free survival
   * Overall survival
2. Safety

   * Frequency and severity of adverse events
   * Frequency of AE requiring discontinuation of study drug or dose reductions

Total sample size:

The planned sample size is 21 patients enrolled at multiple centres in Singapore and South Korea

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible:

* Histologically proven marginal zone lymphoma (splenic, nodal and extra-nodal subtypes included). Patients with clinical and histological evidence of large-cell transformation should be excluded from participating in this study
* Prior treatment with one or more lines rituximab or rituximab-based chemoimmunotherapy with failure to achieve at least a partial response (PR) or documented disease progression
* Age ≥ 21 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* At least 1 measurable disease site on computed tomography (CT) scan that is at least 1.5cm in the longest dimension. Lesions that are not well visualized by CT may be measured by magnetic resonance imaging (MRI) instead
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [β-hCG]) at Screening. Women of childbearing potential are defined as sexually mature women who have not undergone a hysterectomy or bilateral tubal ligation or bilateral oopphorectomy or who have not been naturally postmenopausal for > 2 years
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug. Patient must have an indication for treatment e.g., symptoms from disease, bulky disease (>5cm), threatened end-organ function, or cytopenias requiring transfusion or growth factor support
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study
* Adequate hematological and biochemical parameters within 7 days prior to enrollment as defined below:

Haematological

* Hb ≥8g/dL
* Platelets ≥100,000/mm3 or ≥50,000/mm3 if bone marrow involvement independent of transfusion support in either situation
* Absolute neutrophil count (ANC) ≥1000/mm3 independent of growth factor support

Biochemical

* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN)
* Total bilirubin ≤1.5 x ULN (unless elevated bilirubin is non-hepatic in origin or due to Gilbert's syndrome)
* Serum creatinine ≤2 x ULN or estimate glomerular filtration rate (GFR)(Cockroft Gault) ≥ 40 mL/min/1.73m2

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible

* Prior chemotherapy within 3 weeks, therapeutic anticancer antibodies within 4 weeks, radio or toxin-immunoconjugates within 10 weeks, radiation therapy or other investigational agents within 3 weeks, or major surgery within 4 weeks of first dose of study drug
* Prior treatment with ibrutinib or other BTK inhibitors or PI3K delta inhibitors
* Concurrent enrolment in another therapeutic investigational clinical treatment study
* Prior allogeneic hematopoietic stem cell transplant. Prior autologous hematopoietic stem cell transplant is allowed
* Vaccinated with live, attenuated vaccines within 4 weeks of enrollment
* Known central nervous system lymphoma
* History of prior malignancy, except:

  * Malignancy treated with curative intent and with no known active disease present for ≥3 years before enrollment
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon)
* Requires treatment with strong cytochrome P450(CYP)3A4/5 inhibitors
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrythmias, congestive cardiac failure or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block type II, 3rd degree block, or corrected QT interval (QTc) ≥470 msec
* Known history of Human Immunodeficiency Virus (HIV), or active Hepatitis C or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics
* Pregnant or lactating women
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Overall Response Rates | From time of first study drug administration until best overall response of CR or PR is achieved, up to 3 years
  Proportion of patients who achieve either a Complete Response (CR) or Partial Response (PR) as best response

SECONDARY OUTCOMES:
Progression-Free Survival | From time of first study drug administration until first occurence of disease progression or death from any cause, up to 3 years
Overall Survival | From time of first study drug administration until death from any cause, up to 3 years
Frequency and severity of adverse events | From the time the ICF is signed until 30 days after the last dose of the study drug
Frequency of adverse events requiring discontinuation of study drug or dose reductions | From the time the ICF is signed until 30 days after the last dose of the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany PL Tang, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Cancer Centre Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No